CLINICAL TRIAL: NCT03737032
Title: Theta Burst Stimulation in Young Adults With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erika Forbes (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Erika Forbes, Professor of Psychiatry, Psychology, Pediatrics, & Clinical and Translational Science, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO18040159; R21MH117400 (NIH)
Record Dates: First submitted 2018-10-29; First posted 2018-11-09 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: All participants will receive intermittent Theta Burst Stimulation (TBS), continuous TBS, and sham TBS mimicking stimulation, in randomized, double-blind order across three sessions.
Who Masked: Participant, Outcomes Assessor
Masking Description: The content of each TBS condition will be unknown to participants and to the research staff member conducting assessment of change neural, behavioral, and subjective response with TBS.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Intermittent, Continuous, Sham Order (Experimental): 3 sessions of theta burst stimulation administered in the following order: 1) Intermittent theta burst stimulation, 2) Continuous theta burst stimulation, 3) Sham theta burst stimulation.
  Interventions: Device: Intermittent Theta Burst Stimulation; Device: Continuous Theta Burst Stimulation; Device: Sham Theta Burst Stimulation
- Intermittent, Sham, Continuous Order (Experimental): 3 sessions of theta burst stimulation administered in the following order: 1) Intermittent theta burst stimulation, 2) Sham theta burst stimulation, 3) Continuous theta burst stimulation.
  Interventions: Device: Intermittent Theta Burst Stimulation; Device: Continuous Theta Burst Stimulation; Device: Sham Theta Burst Stimulation
- Continuous, Intermittent, Sham Order (Experimental): 3 sessions of theta burst stimulation administered in the following order: 1) Continuous theta burst stimulation, 2) Intermittent theta burst stimulation, 3) Sham theta burst stimulation.
  Interventions: Device: Intermittent Theta Burst Stimulation; Device: Continuous Theta Burst Stimulation; Device: Sham Theta Burst Stimulation
- Continuous, Sham, Intermittent Order (Experimental): 3 sessions of theta burst stimulation administered in the following order: 1) Continuous theta burst stimulation, 2) Sham theta burst stimulation, 3) Intermittent theta burst stimulation.
  Interventions: Device: Intermittent Theta Burst Stimulation; Device: Continuous Theta Burst Stimulation; Device: Sham Theta Burst Stimulation
- Sham, Intermittent, Continuous Order (Experimental): 3 sessions of theta burst stimulation administered in the following order: 1) Sham theta burst stimulation, 2) Intermittent theta burst stimulation, 3) Continuous theta burst stimulation.
  Interventions: Device: Intermittent Theta Burst Stimulation; Device: Continuous Theta Burst Stimulation; Device: Sham Theta Burst Stimulation
- Sham, Continuous, Intermittent Order (Experimental): 3 sessions of theta burst stimulation administered in the following order: 1) Sham theta burst stimulation, 2) Continuous theta burst stimulation, 3) Intermittent theta burst stimulation.
  Interventions: Device: Intermittent Theta Burst Stimulation; Device: Continuous Theta Burst Stimulation; Device: Sham Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
Device: Continuous Theta Burst Stimulation — Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
Device: Sham Theta Burst Stimulation — For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation. Sham TBS will be delivered with a Cool-B65 Active/Placebo Coil, which includes a sham setting, and MagLink research software.

SUMMARY:
For the proposed 2-year study, the investigators will conduct a within-subject, counterbalanced investigation using functional magnetic resonance imaging (fMRI) and transcranial magnetic stimulation (TMS) to examine the acute effects of theta-burst stimulation (TBS) on function in dorsomedial prefrontal cortex (dmPFC) in 35 young adults with depression (18-25 years, 50% female).

DETAILED DESCRIPTION:
Each participant will undergo 3 sessions of TMS, one each of continuous and intermittent TBS--with the goal of decreasing or increasing dmPFC responding, respectively--and one of sham TBS. Session order will be counterbalanced, with a double-blind approach to condition. Brain function, behavior, and mood will be assessed before and after each TBS session. Broadly, the investigators predict that inhibitory TBS to the dmPFC will enhance neural, behavioral, and subjective aspects of reward function by reducing dmPFC function and dmPFC connectivity with the ventral striatum (VS).

ELIGIBILITY:
Inclusion Criteria:

• DSM-5 Diagnosis of Major Depressive Disorder, Persistent Depressive Disorder (Dysthymia), Other Specified Depressive Disorder, or Other Unspecified Depressive Disorder

Exclusion Criteria:

* Bipolar disorder, substance dependence, or lifetime history of psychosis
* Neurological disorder (e.g., seizure disorder)
* Pregnant
* MRI contradictions: claustrophobia, permanent orthodontic devices, metal implants or other forms of metal in the body that cannot be removed

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika E Forbes, Ph.D., Principal Investigator — The University of Pittsburgh
Locations (1):
- The University of Pittsburgh, Department of Psychiatry, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all individual participant data (IPD) that underlie results in publications that report findings related to tests of our major hypotheses.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available after results of planned tests are published or 5 years after completion of data collection, whichever occurs first. Data will remain available for 5 years.
Access Criteria: We will create procedures for other researchers to request data and will maintain quality assurance of data requests and data sharing. Researchers who share data will be affiliated and in good standing with academic institutions, will have current certification of training in responsible conduct of research, and will complete data requests describing the purpose of the project, the data requested, and the data analysis plan. Requests will be reviewed by the Principal Investigator and, if needed, other members of the research team. Criteria for sharing data will include characteristics described above, as well as scientific merit of the proposed use of data.

REFERENCES:
- [Background] Forbes EE, Dahl RE. Neural systems of positive affect: relevance to understanding child and adolescent depression? Dev Psychopathol. 2005 Summer;17(3):827-50. doi: 10.1017/S095457940505039X. PMID 16262994
- [Background] Damoiseaux JS, Rombouts SA, Barkhof F, Scheltens P, Stam CJ, Smith SM, Beckmann CF. Consistent resting-state networks across healthy subjects. Proc Natl Acad Sci U S A. 2006 Sep 12;103(37):13848-53. doi: 10.1073/pnas.0601417103. Epub 2006 Aug 31. PMID 16945915
- [Background] Downar J, Daskalakis ZJ. New targets for rTMS in depression: a review of convergent evidence. Brain Stimul. 2013 May;6(3):231-40. doi: 10.1016/j.brs.2012.08.006. Epub 2012 Sep 7. PMID 22975030
- [Background] Drysdale AT, Grosenick L, Downar J, Dunlop K, Mansouri F, Meng Y, Fetcho RN, Zebley B, Oathes DJ, Etkin A, Schatzberg AF, Sudheimer K, Keller J, Mayberg HS, Gunning FM, Alexopoulos GS, Fox MD, Pascual-Leone A, Voss HU, Casey BJ, Dubin MJ, Liston C. Resting-state connectivity biomarkers define neurophysiological subtypes of depression. Nat Med. 2017 Jan;23(1):28-38. doi: 10.1038/nm.4246. Epub 2016 Dec 5. PMID 27918562
- [Background] Dunlop K, Gaprielian P, Blumberger D, Daskalakis ZJ, Kennedy SH, Giacobbe P, Downar J. MRI-guided dmPFC-rTMS as a Treatment for Treatment-resistant Major Depressive Disorder. J Vis Exp. 2015 Aug 11;(102):e53129. doi: 10.3791/53129. PMID 26327307
- [Background] Etkin A, Egner T, Kalisch R. Emotional processing in anterior cingulate and medial prefrontal cortex. Trends Cogn Sci. 2011 Feb;15(2):85-93. doi: 10.1016/j.tics.2010.11.004. Epub 2010 Dec 16. PMID 21167765
- [Background] Ferenczi EA, Zalocusky KA, Liston C, Grosenick L, Warden MR, Amatya D, Katovich K, Mehta H, Patenaude B, Ramakrishnan C, Kalanithi P, Etkin A, Knutson B, Glover GH, Deisseroth K. Prefrontal cortical regulation of brainwide circuit dynamics and reward-related behavior. Science. 2016 Jan 1;351(6268):aac9698. doi: 10.1126/science.aac9698. PMID 26722001
- [Background] Forbes EE, Dahl RE. Research Review: altered reward function in adolescent depression: what, when and how? J Child Psychol Psychiatry. 2012 Jan;53(1):3-15. doi: 10.1111/j.1469-7610.2011.02477.x. Epub 2011 Nov 28. PMID 22117893
- [Background] Forbes EE, Hariri AR, Martin SL, Silk JS, Moyles DL, Fisher PM, Brown SM, Ryan ND, Birmaher B, Axelson DA, Dahl RE. Altered striatal activation predicting real-world positive affect in adolescent major depressive disorder. Am J Psychiatry. 2009 Jan;166(1):64-73. doi: 10.1176/appi.ajp.2008.07081336. Epub 2008 Dec 1. PMID 19047324
- [Background] Fox MD, Buckner RL, Liu H, Chakravarty MM, Lozano AM, Pascual-Leone A. Resting-state networks link invasive and noninvasive brain stimulation across diverse psychiatric and neurological diseases. Proc Natl Acad Sci U S A. 2014 Oct 14;111(41):E4367-75. doi: 10.1073/pnas.1405003111. Epub 2014 Sep 29. PMID 25267639
- [Background] Grossheinrich N, Rau A, Pogarell O, Hennig-Fast K, Reinl M, Karch S, Dieler A, Leicht G, Mulert C, Sterr A, Padberg F. Theta burst stimulation of the prefrontal cortex: safety and impact on cognition, mood, and resting electroencephalogram. Biol Psychiatry. 2009 May 1;65(9):778-84. doi: 10.1016/j.biopsych.2008.10.029. Epub 2008 Dec 13. PMID 19070834
- [Background] Haber SN, Knutson B. The reward circuit: linking primate anatomy and human imaging. Neuropsychopharmacology. 2010 Jan;35(1):4-26. doi: 10.1038/npp.2009.129. PMID 19812543
- [Background] Hanlon CA, Dowdle LT, Austelle CW, DeVries W, Mithoefer O, Badran BW, George MS. What goes up, can come down: Novel brain stimulation paradigms may attenuate craving and craving-related neural circuitry in substance dependent individuals. Brain Res. 2015 Dec 2;1628(Pt A):199-209. doi: 10.1016/j.brainres.2015.02.053. Epub 2015 Mar 11. PMID 25770818
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Opie GM, Vosnakis E, Ridding MC, Ziemann U, Semmler JG. Priming theta burst stimulation enhances motor cortex plasticity in young but not old adults. Brain Stimul. 2017 Mar-Apr;10(2):298-304. doi: 10.1016/j.brs.2017.01.003. Epub 2017 Jan 4. PMID 28089653
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Treadway MT, Buckholtz JW, Schwartzman AN, Lambert WE, Zald DH. Worth the 'EEfRT'? The effort expenditure for rewards task as an objective measure of motivation and anhedonia. PLoS One. 2009 Aug 12;4(8):e6598. doi: 10.1371/journal.pone.0006598. PMID 19672310
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Zhang WN, Chang SH, Guo LY, Zhang KL, Wang J. The neural correlates of reward-related processing in major depressive disorder: a meta-analysis of functional magnetic resonance imaging studies. J Affect Disord. 2013 Nov;151(2):531-539. doi: 10.1016/j.jad.2013.06.039. Epub 2013 Jul 12. PMID 23856280
- [Derived] Gupta T, Karim HT, Jones NP, Ferrarelli F, Nance M, Taylor SF, Rogers D, Pogue AM, Seah THS, Phillips ML, Ryan ND, Forbes EE. Continuous theta burst stimulation to dorsomedial prefrontal cortex in young adults with depression: Changes in resting frontostriatal functional connectivity relevant to positive mood. Behav Res Ther. 2024 Mar;174:104493. doi: 10.1016/j.brat.2024.104493. Epub 2024 Feb 7. PMID 38350221

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 participants completed enrollment in the study. Prior to randomization, all 29 participants completed study visit #1 and study visit #2. Out of those 29, 4 participants were withdrawn after study visit #2 and before randomization. 25 participants were randomized and completed the study intervention.
Groups:
- Intermittent, Continuous, Sham Order: 3 sessions of TBS administered in the following order: 1) Intermittent theta burst stimulation, 2) Continuous theta burst stimulation, 3) Sham theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation. Sham TBS will be delivered with a Cool-B65 Active/Placebo Coil, which includes a sham setting, and MagLink research software.
- Intermittent, Sham, Continuous Order: 3 sessions of TBS administered in the following order: 1) Intermittent theta burst stimulation, 2) Sham theta burst stimulation, 3) Continuous theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation. Sham TBS will be delivered with a Cool-B65 Active/Placebo Coil, which includes a sham setting, and MagLink research software.
- Continuous, Intermittent, Sham Order: 3 sessions of TBS administered in the following order: 1) Continuous theta burst stimulation, 2) Intermittent theta burst stimulation, 3) Sham theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation. Sham TBS will be delivered with a Cool-B65 Active/Placebo Coil, which includes a sham setting, and MagLink research software.
- Continuous, Sham, Intermittent Order: 3 sessions of TBS administered in the following order: 1) Continuous theta burst stimulation, 2) Sham theta burst stimulation, 3) Intermittent theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation. Sham TBS will be delivered with a Cool-B65 Active/Placebo Coil, which includes a sham setting, and MagLink research software.
- Sham, Intermittent, Continuous Order: 3 sessions of TBS administered in the following order: 1) Sham theta burst stimulation, 2) Intermittent theta burst stimulation, 3) Continuous theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation. Sham TBS will be delivered with a Cool-B65 Active/Placebo Coil, which includes a sham setting, and MagLink research software.
- Sham, Continuous, Intermittent Order: 3 sessions of TBS administered in the following order: 1) Sham theta burst stimulation, 2) Continuous theta burst stimulation, 3) Intermittent theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation. Sham TBS will be delivered with a Cool-B65 Active/Placebo Coil, which includes a sham setting, and MagLink research software.
Period: Overall Study
Arm/Group | Intermittent, Continuous, Sham Order | Intermittent, Sham, Continuous Order | Continuous, Intermittent, Sham Order | Continuous, Sham, Intermittent Order | Sham, Intermittent, Continuous Order | Sham, Continuous, Intermittent Order
Started | 5 | 4 | 4 | 5 | 4 | 3
Completed | 5 | 4 | 4 | 5 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intermittent, Continuous, Sham Order: 3 sessions of theta burst stimulation administered in the following order: 1) Intermittent theta burst stimulation, 2) Continuous theta burst stimulation, 3) Sham theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation.
- Intermittent, Sham, Continuous Order: 3 sessions of theta burst stimulation administered in the following order: 1) Intermittent theta burst stimulation, 2) Sham theta burst stimulation, 3) Continuous theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation.
- Continuous, Intermittent, Sham Order: 3 sessions of theta burst stimulation administered in the following order: 1) Continuous theta burst stimulation, 2) Intermittent theta burst stimulation, 3) Sham theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation.
- Continuous, Sham, Intermittent Order: 3 sessions of theta burst stimulation administered in the following order: 1) Continuous theta burst stimulation, 2) Sham theta burst stimulation, 3) Intermittent theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation.
- Sham, Intermittent, Continuous Order: 3 sessions of theta burst stimulation administered in the following order: 1) Sham theta burst stimulation, 2) Intermittent theta burst stimulation, 3) Continuous theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation.
- Sham, Continuous, Intermittent Order: 3 sessions of theta burst stimulation administered in the following order: 1) Sham theta burst stimulation, 2) Continuous theta burst stimulation, 3) Intermittent theta burst stimulation.
  Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
  Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
  Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation.
- Total: Total of all reporting groups
Arm/Group | Intermittent, Continuous, Sham Order | Intermittent, Sham, Continuous Order | Continuous, Intermittent, Sham Order | Continuous, Sham, Intermittent Order | Sham, Intermittent, Continuous Order | Sham, Continuous, Intermittent Order | Total
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 4 | 3 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 21 (1.22) | 21 (2.45) | 22 (2.45) | 21.8 (2.39) | 20.25 (2.63) | 21 (1.73) | 21.175 (2.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 2 | 5 | 4 | 3 | 23
  Male | 0 | 0 | 2 | 0 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 4 | 3 | 3 | 5 | 4 | 3 | 22
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 1 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 0 | 0 | 3
  White | 2 | 2 | 3 | 4 | 3 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 5 | 4 | 3 | 25

OUTCOME MEASURES:

1. Primary Outcome: Dorsomedial Prefrontal Cortex Activation
Description: This measure captures brain function in the dorsomedial prefrontal cortex (dmPFC) based on blood oxygen level dependent (BOLD) response measured using functional magnetic resonance imaging (fMRI) during a reward task. Data are analyzed using Statistical Parametric Mapping. Magnitude of dmPFC response is in arbitrary units, with higher values reflecting higher activation. Theoretical minimum and maximum scores do not exist. Study hypotheses predict that dmPFC will decrease (based on statistical significance) with continuous TBS.
Time Frame: Task fMRI is conducted after each of 3 TBS sessions (intermittent, continuous, sham; in randomized, counterbalanced order) at approx 3, 5, and 7 weeks after study entry.
Population: Cases included in analysis are those from participants who completed all study procedures (i.e., all TMS sessions, all MRI scans), had available data, and passed data quality criteria
Measure: Mean (Standard Deviation); unit: score in arbitrary units
Groups:
- Intermittent TBS: intermittent theta burst stimulation
  This was 1 of 3 conditions used and was an active condition. All participants were intended to receive all 3 conditions, but order of condition was randomized.
- Continuous TBS: continuous theta burst stimulation
  This was 1 of 3 conditions used and was an active condition. All participants were intended to receive all 3 conditions, but order of condition was randomized.
- Sham TBS: sham theta burst stimulation
  This was one of 3 conditions used and was a non-active condition. All participants were intended to receive all 3 conditions, but order of condition was randomized.
Arm/Group | Intermittent TBS | Continuous TBS | Sham TBS
Number analyzed (Participants) | 10 | 10 | 10
score in arbitrary units | 0.16 (3.79) | 1.35 (4.30) | 0.36 (3.60)
Statistical Analysis 1: Comparison: Intermittent TBS vs Continuous TBS vs Sham TBS; Null hypothesis: post-TBS dmPFC activation will not vary by TBS condition. This is tested using the main effect of condition in a repeated measures model; Test type: Superiority; p = 0.80, ANOVA

2. Secondary Outcome: Positive Affect
Description: Self-reported pleasant mood was measured with the Positive Affect (PA) scale of the Positive and Negative Affect Schedule (PANAS). This scale consists of a number of words that describe different feelings and emotions, participants are instructed to read each item and then mark to which extent they have felt like this in the past few hours. The PA scale contains 10 items, with each item rated on a 5-point scale of 1 (very slightly or not at all), 2 (a little), 3 (moderately), 4 (quite a bit), or 5 (extremely). Higher scores indicate greater PA. The total PA score is calculated by finding the sum of the 10 positive items. Scores range from 10-50. A higher score indicates higher intensity of positive affect. The PANAS PA data analyzed were from administrations pre- and post-TBS at visits #3-5 (approximately 30 minutes before and 1 hour after TBS administration).
Time Frame: pre and post each of 3 TBS administrations, with TBS lasting up to 190 seconds. cTBS, iTBS, and sham TBS each occurred in a single day.
Population: Only participants who completed the PA measure at all time points (pre/post each condition, all 3 conditions) were included in analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intermittent TBS | Continuous TBS | Sham TBS
Number analyzed (Participants) | 20 | 20 | 20
score on a scale
  Pre | 20.70 (6.74) | 20.05 (6.24) | 20.45 (6.06)
  Post | 20.45 (7.35) | 19.80 (7.80) | 22.10 (9.71)
Statistical Analysis 1: Comparison: Intermittent TBS vs Continuous TBS vs Sham TBS; Null hypothesis: pre-post change in positive affect will not vary by TBS condition. This is tested using the interaction of time*condition in a repeated measures model; Test type: Superiority; p = 0.23, ANOVA; Repeated measures ANOVA with time (pre or post), condition (cTBS, iTBS, sham TBS), and time*condition effects

3. Secondary Outcome: VS-dmPFC Functional Connectivity
Description: Outcome measure is assessed with functional magnetic resonance imaging (fMRI), in which brain function is recorded during a reward task. Functional connectivity between 2 regions of neural reward circuitry, the ventral striatum (VS) and the dorsomedial prefrontal cortex (dmPFC), is computed using general psychophysiologic interaction for this pair of regions in Statistical Parametric Mapping software. FC data are in arbitrary units, with higher values reflecting higher degree of coordination between the regions. Theoretical minimum and maximum scores do not exist. Higher scores do not represent "better" or "worse" outcomes or change in health. Based on study hypotheses, FC is predicted to decrease with continuous TBS, based on significance of statistical tests.
Time Frame: Task fMRI is conducted after each of 3 TBS sessions (intermittent, continuous, sham; in randomized, counterbalanced order). Sessions occur at approx 3, 5, and 7 weeks after study entry.
Population: Cases included in analysis are those from participants who completed all MRI scans, had available fMRI data, and had data that passed quality criteria
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Intermittent TBS | Continuous TBS | Sham TBS
Number analyzed (Participants) | 10 | 10 | 10
arbitrary units | 2.28 (7.64) | 4.10 (13.70) | 1.16 (5.61)
Statistical Analysis 1: Comparison: Intermittent TBS vs Continuous TBS vs Sham TBS; Null hypothesis: post-TBS functional connectivity between the dmPFC and ventral striatum (VS) will not vary by TBS condition. This is tested using the main effect of condition in a repeated measures model; Test type: Superiority; p = 0.84, ANOVA

ADVERSE EVENTS:
Time Frame: The duration of the study per person was generally up to 10 weeks.
Groups:
- Intermittent: Intermittent Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered without interruption for a total duration of 40 seconds.
- Sham: Sham Theta Burst Stimulation: For the sham of theta burst stimulation, the device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation. Sham TBS will be delivered with a Cool-B65 Active/Placebo Coil, which includes a sham setting, and MagLink research software.
- Continuous: Continuous Theta Burst Stimulation: Theta Burst Stimulation, a form of Transcranial Magnetic Stimulation, will be applied to the dorsomedial prefrontal cortex. will include 600 pulses delivered in brief bursts of three pulses with a frequency of 50 Hz, at an intensity of 110% of resting motor threshold, and administered every 200 ms (5 Hz). Bursts will be delivered during 2 second periods (10 bursts/period) interleaved with 8-second stimulation-free intervals, for a total duration of 190 seconds.
Arm/Group | Intermittent | Sham | Continuous
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent (N=25) | Sham (N=25) | Continuous (N=25)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT03737032/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT03737032/ICF_001.pdf